CLINICAL TRIAL: NCT03989635
Title: Randomized, Subject and Investigator Blinded, Placebo-controlled Study to Demonstrate the Anti-inflammatory Effect of Fevipiprant (QAW039) in Moderate to Severe Asthma Patients With High Sputum and Blood Eosinophils.
Brief Title: Mechanistic Study of Anti-inflammatory Effects of Fevipiprant in Patients With Eosinophilic Asthma.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAW039A2127
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Asthma; Asthma, Bronchial; Bronchial Asthma; Eosinophilia; Physiological Effects of Drugs
Keywords: QAW039; Asthma; Sputum; Eosinophilia; eosinophillic; Prostaglandin D2 receptor; DP2; Fevipiprant.
MeSH Terms: conditions — Asthma; Eosinophilia | interventions — fevipiprant

STUDY DESIGN:
Intervention Model Description: This is a non-confirmatory, mode-of-action, placebo-controlled, parallel group, randomized, subject and investigator blinded study in 48 moderate to severe asthma patients, who are on at least medium dose ICS, with or without other asthma controller and with elevated sputum eosinophils count of ≥ 2% of the total cell count from an induced sputum specimen and a peripheral eosinophil count ≥ 250 cells/μL of blood. They should be on standard of care asthma medications for 4 weeks prior to screening with no past or current medical history of other chronic or severe pulmonary diseases. Randomized patients will be treated with fevipiprant or matching placebo for up to 98 days. A group of 10 healthy subjects will also be recruited to examine baseline levels of prostaglandins and DP2-related biomarkers and compare them to biomarker data from asthma patients at baseline and after therapy with fevipiprant.
  Healthy volunteers will not receive study treatment.
  .
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a subject and investigator-blinded study. Subjects, investigators and all site staff will remain blinded to study treatment throughout the study.
  Unblinding a single subject at site for safety reasons (if necessary for subject management) will occur via an emergency system in place at the site.
  The identity of the treatments will be concealed by the use of study drugs that are all identical in packaging, labeling, schedule of administration, appearance, and odor.
  The sponsor may be unblinded to the study treatment at any time, especially in case of a safety concern.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QAW039 (Experimental): QAW039 450mg
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo to QAW039
  Interventions: Drug: QAW039

INTERVENTIONS:
Drug: QAW039 — QAW039 450mg
  Other Names: Fevipiprant

SUMMARY:
This is an exploratory, randomized, subject- and investigator-blinded, placebo-controlled mode-of-action study to demonstrate the anti-inflammatory effects of fevipiprant compared to placebo after 12 weeks of treatment in 48 moderate to severe asthma patients with sputum and blood eosinophilia.

DETAILED DESCRIPTION:
The main purpose of this study is to demonstrate the anti-inflammatory effects of fevipiprant (QAW039) compared to placebo after 12 weeks of treatment in moderate to severe asthma patients with an elevated sputum eosinophil count (≥ 2%) and high blood eosinophil count (≥ 250 cells/μL). This study is also designed to investigate the effects of fevipiprant on key inflammatory cells bearing the DP2 receptor (such as eosinophils, Th2/Tc2 cells, and ILC2 cells) in sputum and blood.

ELIGIBILITY:
Inclusion Criteria:

All Subjects (Asthma patients and healthy volunteers):

* Written informed consent must be obtained before any assessment is performed.
* Male and female subjects aged ≥ 18 years.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Asthma patients:

* Patients with a diagnosis of asthma currently prescribed at least medium dose of ICS, alone or with any other asthma controller therapy, except those listed as prohibited medications. Patients must be on stable doses of asthma medications for at least 4 weeks prior to screening.
* A clinical diagnosis of asthma supported by at least one of the following within the last five years
* Reversible airway obstruction defined as an increase of ≥ 12% and ≥ 200 ml in FEV1 or FVC over the patient's pre-bronchodilator value within 30 minutes after inhaling a total of 360 μg of albuterol or 400 μg salbutamol via metered dose inhaler (reversibility test)
* A positive airway hyper-reactivity (AHR) test result defined as a provoked fall in FEV1 of 20% (PC20) by methacholine at ≤ 8 mg/ml when not on ICS or ≤ 16 mg/ml on ICS therapy
* A change in FEV1 of ≥ 12% over two measurements within 12 months.
* ACQ7 score ≥ 1.25 at screening and baseline visits and may be repeated once at each visit.
* Demonstrate ability to produce a good quality induced-sputum sample at baseline visit.
* Sputum eosinophil count ≥ 2% and blood eosinophil count ≥ 250cells/μL at applicable screening and baseline visits.

Healthy volunteers:

* Subject must be in good health as determined by past medical history, current medications, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Subjects with well-controlled, mild, non-respiratory diseases can participate as long as they are considered healthy and stable in the investigator's judgement.

Exclusion Criteria:

All Subjects (Asthma patients and healthy volunteers):

* Use of other investigational drugs at the time of screening, or within 5 half-lives of experimental drug at the time of screening, or within 30 days of last dose of experimental drug at the time of screening, whichever is longer; or longer if required by local regulations.
* A positive human immunodeficiency virus test or is taking anti-retroviral medications, as determined by medical history and/or subject's verbal report.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Donation or loss of 450 mL or more of blood within eight weeks prior to screening visit or longer if required by local regulation.
* Pregnant or nursing (lactating) women.

Asthma patients:

* Patients with a current or past medical history of conditions other than asthma or allergic rhinitis that could result in elevated blood or sputum eosinophils (e.g., hypereosinophilic syndrome, Churg-Strauss Syndrome).
* History of hypersensitivity to any of the study treatments or excipients (such as milk or lactose) or to drugs of similar chemical classes (other DP2 antagonists such as timapiprant).
* Patients with history of concomitant chronic or severe pulmonary disease other than asthma (e.g., COPD, bronchiectasis, sarcoidosis, interstitial lung disease, cystic fibrosis, active tuberculosis).
* Use of biologic therapy for asthma (e.g. omalizumab, mepolizumab, benralizumab, dupilumab) within 3 months or 5 half-lives prior to screening, whichever is longer.
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for subjects participating in the study such as:
* Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and second or third degree AV block without a pacemaker
* History of familial long QT syndrome or known family history of Torsades de Point Resting QTcF (Fredericia) ≥ 450 msec (male) or ≥ 460 msec (female) at screening
* Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of study.
* Patients on statin therapy with a CK level >2 X ULN at screening.
* Patients who have a clinically significant laboratory abnormality at screening including but not limited to:
* Total white blood cell count < 2500 cells/μL
* AST or ALT > 2.0 X ULN or total bilirubin > 1.3 X ULN
* Estimated Glomerular Filtration Rate (eGFR) by the Modification of Diet in Renal Disease (MDRD) equation < 55 mL/minute/1.73m2.

Healthy volunteers:

* History of allergies or atopy (e.g., allergic rhinitis, urticaria, eczematous dermatitis).
* Recent (within the last three years) and/or recurrent history of acute or chronic obstructive disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* Use of any prescription drugs, herbal supplements, prescribed medicinal use of cannabis/marijuana, within four weeks prior to screening assessments, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two weeks prior to screening. If needed, (i.e. an incidental and limited need) paracetamol/acetaminophen is acceptable, but must be documented in the Concomitant medications / Significant non-drug therapies page of the CRF.
* Significant illness, which has not resolved within two weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-06-14 (Estimated)

PRIMARY OUTCOMES:
Sputum eosinophil % of total cell count | 12 weeks
  To assess the change from baseline in
  sputum eosinophil levels after 12 weeks of treatment with fevipiprant compared to placebo in moderate to severe asthma patients with sputum and blood eosinophilia.

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com